CLINICAL TRIAL: NCT02502123
Title: Multi-Centre, Prospective, Observational Study of Patient Reported Outcomes in Patients Diagnosed With Chronic Migraine and Treated With OnabotulinumtoxinA for Injection (BOTOX®) (PREDICT)
Brief Title: Patient Reported Outcomes in Patients With Chronic Migraine Treated With BOTOX®
Acronym: PREDICT
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: GMA-CAN-NEU-0336
Record Dates: First submitted 2015-07-16; First posted 2015-07-20 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OnabotulinumtoxinA (BOTOX®): Patients diagnosed with chronic migraine headache treated with BOTOX® as standard of care in clinical practice. No intervention was administered in this study.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No intervention was administered in this study.

SUMMARY:
This study will prospectively assess long term heath related quality of life in chronic migraine patients currently being treated with OnabotulinumtoxinA for injection (BOTOX®) as standard of care.

ELIGIBILITY:
Inclusion Criteria:

-Patients with chronic migraine eligible to receive treatment with onabotulinumtoxinA (BOTOX®) as standard of care.

Exclusion Criteria:

* Diagnosis of hemiplegic migraine, basilar migraine, ophthalmoplegic migraine or migrainous infarction, chronic tension-type headache, hypnic headache, hemicrania continua or new daily persistent headache.
* Patient who is currently taking or planning on taking opioid-containing products, barbiturates or combination for acute headache or pain condition.
* Treatment with any other botulinum toxin product for any condition within 3 months of the screening visit.
* Diagnosis of myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis or any other significant disease that might interfere with neuromuscular function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic migraine treated with BOTOX® as standard of care.
Sampling Method: Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2015-07-02 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-01-29 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Migraine-Specific Quality of Life (MSQ) at Treatment 4 Using a 6-Item Questionnaire | Baseline, Treatment 4 (approximately 24 Weeks)

SECONDARY OUTCOMES:
Change from Baseline in MSQ at Final Visit Using a 6-Item Questionnaire | Baseline, Final Visit (Up to 2 Years)
Clinician's Global Impression of Change Using a 7-Point Scale | Up to 2 Years
Healthcare Resource Utilization Before and After BOTOX® using a 9-Item Questionnaire | Baseline, Up to 2 Years
BOTOX® Treatment Regimen for Chronic Migraine | Up to 2 Years
Work Productivity and Activity Impairment Questionnaire: Specific Health Problem Before and After BOTOX® Consisting of 6-Items | Baseline, Up to 2 Years
Patient Global Assessment of Treatment Satisfaction with BOTOX® using a 3-Item Questionnaire | 2 Years
Change from Baseline in Beck Depression Inventory Scale at Final Visit Using a 21-Item Questionnaire | Baseline, Final Visit (Up to 2 Years)
Reasons Why Treatment with BOTOX® Stopped | Up to 2 Years
Headache Assessment from Patient Diary | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Goran Davidoic, Study Director — Allergan
Locations (15):
- Canada (15):
  - Foothills Medical Centre, Calgary, Alberta
  - Hys Medical Centre, Edmonton, Alberta
  - Bayside Medical Centre, Brentwood Bay, British Columbia
  - Jeff Oyler, Kamloops, British Columbia
  - Dhawan Medical Corporation Medical Clinic, Vancouver, British Columbia
  - May Ong-Lam, Vancouver, British Columbia
  - Island Neurology, Victoria, British Columbia
  - Hamilton Headache Clinic, Hamilton, Ontario
  - The Shapero Markham Headache and Pain Treatment Centre, Markham, Ontario
  - Pain Care Clinics, Mississauga, Ontario
  - Toronto Headache & Pain Centre, North York, Ontario
  - Hany Demian, Oakville, Ontario
  - Nepean Medical Centre, Ottawa, Ontario
  - Centre de traitement neurologique, Monthreal, Quebec
  - Clinic Greene Avenue, Montreal, Quebec